CLINICAL TRIAL: NCT03770793
Title: Effectiveness of Ultrasound-guided Alveolar Recruitment in Thoracic Surgery With One-lung Ventilation
Brief Title: Effectiveness of Lung Sono in One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JHSeo_LungSono
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: One Lung Ventilation
Keywords: One lung ventilation; Lung ultrasound; Alveolar recruitment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung-sono guided (Experimental): Before starting one-lung ventilation, alveolar recruitment is performed under the examination with ultrasound. Find the minimal airway pressure that actually starts to resolve the observed atelectasis. Repeat alveolar recruitment with the minimal pressure untill the atlelectasis is not visible.
  Interventions: Procedure: Lung-sono guided
- Conventional (No Intervention): Before starting one-lung ventilation, alveolar recruitment is performed with the pressure of 30mmHg for 10 seconds which is a conventional method.

INTERVENTIONS:
Procedure: Lung-sono guided — The patient undergoing thoracic surgery is intubated with double lumen tube after induction of general anesthesia with propofol and remifentanil.
  In the intervention group, alveolar recruitment is performed to the non-surgical side of lung under examination with ultrasound just after anesthesia induction.
  During the gradual increment in the pressure of recruitment, the anesthesiologist can find the opening pressure that means the minimal pressure at which observed atelectasis starts to disappear.
  Then, alveolar recruitment is performed with the opening pressure until the atelectasis is not visible.
  Arms: Lung-sono guided

SUMMARY:
To observe the effectiveness of ultrasound-guided alveolar recruitment in thoracic surgery with one-lung ventilation(OLV).

DETAILED DESCRIPTION:
One-lung ventilation(OLV) is essential in thoracic surgery for patient safety and better surgical view. However, pulmonary complications such as hypoxemia may be caused by OLV which might be preventable with adequate alveolar recruitment and positive end-expiratory pressure(PEEP). Alveolar recruitment has been performed with conventional methods without diagnostic tools in clinical setting.

Ultrasound is a non-invasive, radiation-free device with high accuracy for the diagnosis of lung atelectasis. There are a few reports regarding the usefulness of lung ultrasound in other surgeries, but not in thoracic surgeries with OLV.

Thus, investigators designed a study to observe the effectiveness of ultrasound-guided alveolar recruitment in thoracic surgery with OLV.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracic surgery which requires one-lung ventilation with lateral decubitus position

Exclusion Criteria:

* Patients who refuse to agree
* Previous lung surgical history
* History of pneumothorax or bullae
* Severe cardiopulmonary disease, COPD
* Operation time < 1hr

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of desaturation | intraoperative
  SpO2<95%
P/F ratio | 30 minutes after one-lung ventilation
  PaO2/FiO2 ratio

SECONDARY OUTCOMES:
Lung ultrasound score | just after anesthesia induction, end of surgery
  Lung ultrasound score of atelectasis
Alveolar dead space | 30 minutes after one-lung ventilation
  (PaCO2-PetCO2)xVt/PaCO2
Pulmonary complications | intraoperative, during hospital stay(an average of 3 days)
  respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, atelectasis, bronchospasm, aspiration pneumonitis

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Song IK, Kim EH, Lee JH, Kang P, Kim HS, Kim JT. Utility of Perioperative Lung Ultrasound in Pediatric Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2018 Apr;128(4):718-727. doi: 10.1097/ALN.0000000000002069. PMID 29309282
- [Derived] Kim BR, Lim L, You J, Yoon S, Park JB, Bahk JH, Seo JH. Effectiveness of ultrasound-guided alveolar recruitment in thoracic surgery with one-lung ventilation: a randomized-controlled trial. Eur J Cardiothorac Surg. 2025 Jul 1;67(7):ezaf204. doi: 10.1093/ejcts/ezaf204. PMID 40581064